CLINICAL TRIAL: NCT05825053
Title: The Effect of Single Booster Sessions or Home-based Exercise Program for Individuals in the Chronic Phase After Stroke to Retain Short-term Training Effects on Gait Adaptability, a Study-protocol.
Brief Title: Retaining Short-term Training Effects on Gait Adaptability in People With Stroke
Acronym: ATTAINS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sint Maartenskliniek (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL80178.091.21 / 0996_2
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Booster group (Experimental): Participants assigned to the booster group will receive a three single training sessions 3 months apart targeting gait adaptability using the C-mill. Assessments will take place after giving informed consent which is indicated as the start of the study (baseline), 6 months and 12 months post-baseline.
  Interventions: Behavioral: Gait adaptability training
- Home-based exercise group (Experimental): Participants assigned to the home-based exercise group will receive a program for training at home aiming at a minimum training time of 60 minutes per week. Assessments will take place after giving informed consent which is indicated as the start of the study (baseline), 6 months and 12 months post-baseline
  Interventions: Behavioral: Home-based exercise training
- Control group (No Intervention): Participants assigned to the control group will not follow any additional intervention other than the standard care they already receive for the year following the completion of the 5-week gait adaptability training using the C-Mill from the ATTAINS study. Assessments will take place after giving informed consent which is indicated as the start of the study(baseline), 6 months and 12 months post-baseline.

INTERVENTIONS:
Behavioral: Gait adaptability training — Over a span of 1 year participants will receive 3 one hour, single sessions at 3, 6 and 9 months following baseline assessment, of gait adaptability training, using the C-mill (an instrumented treadmill with augmented reality). Several aspects of gait adaptability, such as obstacle avoidance, accelerating/decelerating and precision stepping, will be trained.
  Arms: Booster group
Behavioral: Home-based exercise training — Participants will receive tailored exercise through an online platform targeting gait adaptability. Participants are instructed to train at a minimum of 60 minutes per week, with a frequency of 2 sessions per week. Participants will be supported through tele-consultations on a monthly basis for the first 3 months and bi-monthly for the remaining time of the study. These consultations are focused on technical support, on ways to ensure training progression and to encourage adherence to the program.
  Arms: Home-based exercise group

SUMMARY:
Background: The majority of stroke survivors regain walking ability. However, the ability to adapt gait patterns to meet environmental demands remains impaired in a majority of people in the chronic phase after stroke. This impaired gait adaptability has a profound impact on activities of daily living and quality of life. Treatment targeting gait adaptability is therefore critical for safe and independent community ambulation in people with stroke. Augmented or virtual reality in rehabilitation programs can be used to train gait adaptability in a controlled situation. A few studies have evaluated gait adaptability training in people with stroke. Although results were promising, these studies did not include an adaptability-related outcome measure, or were limited to uncontrolled or small-scaled pilot studies. Moreover, it is unknown if beneficial training effects can be fostered for 1 year after completion of a training program. We evaluate the short-term effects of a 5-week gait adaptability training in an adequately powered, waiting-list controlled clinical trial [ref naar clin trial nummer]. In the current study, we focus on the retention of potentially beneficial effects of this 5 week gait adaptability training program. We will evaluate if short-term effects of gait adaptability training can be retained through single training sessions to boost performance, or by an home exercise program. We hypothesize that booster sessions and home-based exercise will both yield better retention of training effects at 1 year follow-up as compared to the control arm without an experimental intervention.

Objective: The primary objective of this study is to test the hypothesis that retention of training-induced gains in gait adaptability can be fostered by providing booster sessions or by prescribing home-based training.

Study design: Explorative randomized study, comparing the effect of 3 1-hr booster training sessions against home-based exercise against no intervention on gait adaptability performance 1 year after completion of a 5-week gait adaptability training program.

Study population: Stroke patients in the chronic phase after stroke, who completed the 5-week gait adaptability training using the C-Mill and agreed to continue in this follow-up study. We expect this to be 50-75 participants.

ELIGIBILITY:
Inclusion Criteria:

* > 6 months after first unilateral supratentorial stroke (chronic phase)
* Able to walk at least 10 minutes independently
* Initial involvement of the lower extremity after stroke.
* Having completed (minimal 8/10 training sessions) the 5 week gait adaptability training program using the C-Mill

Exclusion Criteria:

* Any other neurological or musculoskeletal disease affecting gait or balance (e.g. Parkinson's disease, knee osteoarthritis)
* Contractures or spasticity requiring other treatment (e.g. botulinum toxin treatment) within the duration of the training period.
* Severe cognitive or visuo-spatial impairments limiting comprehension of instructions or correct perception of the environments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Walking Adaptability Ladder Test (WALT) score | 12 months post-baseline
  Measure of gait adaptability. An adapted version for adults of the Walking Adaptability Laddertest for Kids (WAL-K) to assess the ability to flexibly adjust the gait pattern during overground walking. Outcome is based on performance time and foot placement errors measured in seconds where a lower score is a better outcome.
Emory Functional Ambulation Profile (EFAP) score | 12 months post-baseline
  Measure of gait adaptability. In this task the participants traverse a standardized 5m obstacle course. Outcome is time to perform the task measured in seconds where a lower score is a better outcome

SECONDARY OUTCOMES:
Lab-based walking adaptability test | 12 months post-baseline
  Measure of gait adaptability. Target stepping task using the Gait Real-time Analysis Interactive Lab (GRAIL) where participant must step on projected stepping stones as accurately as possible. Step width and step length between the stepping stones will vary.
Balance performance | 12 months post-baseline
  Measure of gait stability, measured by the margin of stability (meter) and the center of mass excursion (meter), on treadmill walking with perturbations using the Gait Real-time Analysis Interactive Lab (GRAIL).
Walking performance | 12 months post-baseline
  Measure of walking ability using the 10meter walktest, measured in seconds where a lower score is a better outcome.
Balance confidence | 12 months post-baseline
  Evaluating balance confidence using the Activity Balance Scale, measured on a 0% - 100% scale, where a higher score is a better outcome.
Daily life gait performance as assessed by gait quality | 12 months post-baseline
  Measured by inertial measurement units placed on both feet and the lower back. Analysis through cusomized algorythms.
Daily life walking activity assessed by walking time per day | 12 months post-baseline
  Average time of walking during the day (minutes) measured in one week using the Activ8.
Health-related quality of life | 12 months post-baseline
  Evaluating the disability and health-related quality of life after stroke using the Stroke Impact Scale mobility subscale, measure on a 5-point scale ("could not do at all = 1" - "not difficult at all = 5") where a higher score is a better outcome.
Balance performance through MiniBESTest | 12 months post-baseline
  Measure of balance and gait stability using the Mini Balance Evaluation Systems Test (MiniBESTes). Tasks are score on a 3-point scale. Outcome is an average score ranging between 0 and 1 where a higher score is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Weerdesteyn, Prof. dr., Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Ubbergen, Netherlands

REFERENCES:
- [Background] Kuijpers R, Smulders E, Groen BE, Smits-Engelsman BCM, Nijhuis-Van der Sanden MWG, Weerdesteyn V. Reliability and construct validity of the Walking Adaptability Ladder Test for Kids (WAL-K): a new clinical test for measuring walking adaptability in children. Disabil Rehabil. 2022 Apr;44(8):1489-1497. doi: 10.1080/09638288.2020.1802523. Epub 2020 Aug 10. PMID 32776854
- [Background] Tuijtelaars J, Roerdink M, Raijmakers B, Nollet F, Brehm MA. Polio survivors have poorer walking adaptability than healthy individuals. Gait Posture. 2021 Jun;87:143-148. doi: 10.1016/j.gaitpost.2021.04.031. Epub 2021 Apr 21. PMID 33915437
- See also: The English description of the project on the website of the Sint Maartenskliniek. — https://www.maartenskliniek.nl/research-innovation-en/research-innovation-projects/attains-gait-adaptability-training-for-people-after-stroke